CLINICAL TRIAL: NCT05772598
Title: A Cohort Study Comparing the Novel 'Sexual Minorities and Prostate Cancer Scale' to the Gold Standard Questionnaires Investigating Erectile Dysfunction and Incontinence Following Robotic Assisted Radical Prostatectomy
Brief Title: Validating the 'Sexual Minorities and Prostate Cancer Scale' to Gold Standard Questionnaires
Acronym: SMACS
Status: Completed | Type: Observational
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 305757
Record Dates: First submitted 2022-09-06; First posted 2023-03-16 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2022-09

CONDITIONS: Prostate Cancer; Incontinence; Erectile Dysfunction Following Radical Prostatectomy
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A cohort study comparing the novel 'Sexual Minorities and Prostate Cancer Scale' (SMACS) to the gold standard questionnaires investigating erectile dysfunction (IIEF) and incontinence (ICIQLUTSqol and ICIQ-UI) following robotic assisted radical prostatectomy

DETAILED DESCRIPTION:
Prostate cancer treatments negatively impact sexual and urinary function. Prostate cancer is increasing in incidence and through rapid uptake of the screening tool, PSA, many patients are getting diagnosed younger and with lower risk disease. With this shift, cancer survivorship both in its assessment and management, is becoming a growing issue as more patients live with the after effect of prostate cancer treatments. Many tools have been developed to assess sexual and urinary function following treatments such as the Expanded Prostate Cancer Index (EPIC), ICIQLUTSqol or the International Index of Erectile Function (IIEF). However, these do not capture the experience of gay, bisexual and transsexual (sexual minority) patients.

In previous studies of heterosexual prostate cancer patients, erectile dysfunction was reported in 51-60% after 24 months post-treatment and urinary incontinence 7-14% at 24 months. Whilst there is common ground in the obstacle for sexual recovery following surgery, sexual minority patients face additional challenges including erections that are too weak for anal insertive sex [], loss of ejaculate (which is a central to many sexual minority men) [], arousal incontinence and climacturia during oral sex [] or the potential loss of sexual pleasure in receptive anal sex []. In a recent study of 193 sexual minority prostate cancer patients, only 12% described their overall sexual functioning as 'very good' or 'excellent'.

In a review of twelve common sexual functioning scales in prostate cancer survivors [], all focused primarily or exclusively on erectile function and seven explicitly defined intercourse as vaginal penetration. Thus, existing measures used in clinical research and practice may lack validity in measuring quality of life among sexual minority patients. This not only fails to consider these aspects in the sexual minority survival of cancer but also under reports the scale of the problem in the literature.

Radical prostatectomy is a main treatment for low-intermediate risk prostate cancer and at Guy's and St Thomas's, surgeons undertake around 300/year. The investigators follow these patients up with IIEF at 3, 6, 12 and 24 months following their surgery as standard.

The Restore Group, has developed the Sexual Minorities and Prostate Cancer Scale (SMACS). This study used 401 sexual minority patients whom completed an online battery of urinary and sexual functioning including a new 37-item instrument about their sexual functioning post treatment for prostate cancer. Confirmatory factor analysis was used to determine the construct validity with three subscales revealed: sexual distress, urinary incontinence in sex and problematic receptive anal sex. Cronbach's alphas ranged 0.86-0.93. For criterion validity, sexual distress correlated strongly with EPIC sexual function and bother scores. Urinary incontinence in sex correlated weakly with EPIC sexual function and bother (r=0.10-0.19). Problematic receptive anal sex was weakly correlated with each EPIC scale (r=0.12-0.29).

Whilst it is important to develop a tool that properly addresses sexual minority patients' sexual and urinary dysfunction. The goal moving forward should be an inclusive questionnaire that can be used no matter their sexual preference. This study aims to address this by validating this new questionnaire in our post-prostatectomy cohort that will consist of sexual majority and minority patients.

ELIGIBILITY:
Inclusion Criteria:

* All patients attending for prostatectomy care at our institution

Exclusion Criteria:

* All non-English speakers

Ages: 40 Years to 75 Years | Sex: Male
Age Groups: Adult, Older Adult
Study Population: Patients treated with prostatectomy for prostate cancer
Sampling Method: Non-Probability Sample
Enrollment: 305 (Actual)
Dates: Start 2023-03-15 (Actual); Primary Completion 2023-08-02 (Actual); Study Completion 2023-08-02 (Actual)

PRIMARY OUTCOMES:
The score for SMACS domains for sexual dysfunction compared to gold standard PROM for erectile function (IIEF) in a post-prostatectomy population | 10 months
  At a single timepoint, sexual dysfunction measured using SMACS scale and International Index of Erectile Function.
The score for SMACS domains for incontinence compared to two gold standard PROMs for incontinence (ICIQLUTSqol, ICIQ-UI) in a post-prostatectomy population | 10 months
  At a single timepoint, incontinence will be measured using SMACS scale and International Consultation on Incontinence Questionnaires: LUTSqol and ICIQ-UI.

SECONDARY OUTCOMES:
Acceptability questionnaire of the SMACS questionnaire | 10 months
  Acceptability and ease of use will be measured by a Likert scale 7 point questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Guys and St Thomas' NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No